CLINICAL TRIAL: NCT04484389
Title: Effects of Exercise With Telerehabilitation on Depression, Quality of Life and Fatigue in Individuals With Chronic Disease
Brief Title: Telerehabilitation in Individuals With Chronic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Sevval Bakir, Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 015
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Telerehabilitation
Keywords: Chronic Disease; Exercises; Social Isolation
MeSH Terms: conditions — Chronic Disease; Motor Activity; Social Isolation | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Individual exercises will be applied to individuals with Chronic disease.
  Interventions: Other: Telerehabilitation
- Control Group (Active Comparator): Group to be given an exercise brochure
  Interventions: Other: Exercise brochure

INTERVENTIONS:
Other: Telerehabilitation — Exercise protocol according to Ipaq will be prepared for 30 patients with chronic disease . Exercise protocol; warm-up exercises include, stretching exercises, postural exercises, aerobic exercise and cooling exercises. People will practice the exercises 3 days a week for 6 weeks. People will need to reserve 30 minutes a day for this study.
  Arms: Study Group
Other: Exercise brochure — General exercise protocol will be prepared and given to the control group as a brochure
  Arms: Control Group

SUMMARY:
Telerehabilitation applications are a treatment method that uses new technologies. There are examples of doing for many diseases in our country. It is a method used for people living in remote areas and people who cannot complete their treatment in hospitals due to the epidemic. In our study, we will use the telerehabilitation system. In this system, which we will use in people with chronic disease, we aim to see improvement in tests performed in many areas such as physical activity level, respiratory capacity, depression, and anxiety level of patients.

In the study to be performed on 60 patients, 30 people will be control and 30 people will be the experimental group. The experimental group will be treated with a video conferencing method, tailor-made exercise program based on the international physical activity questionnaire level for 30 minutes 3 days a week for 6 weeks. The control group will only be informed with the help of a brochure with a standard exercise program.

The tests we can use in this experiment are as follows: Barthel daily life activities index, beck depression and anxiety scale, ferrans power quality of life index, Charlson comorbidity index, environmental measurements, waist/hip ratio, fatigue severity scale, international physical activity questionnaire. Tests specific to chronic diseases will be applied to patient one to one.

ELIGIBILITY:
Inclusion Criteria:

* Having a chronic disease
* To be able to communicate verbally
* Being in a stable period in terms of disease
* At least 3 months for the disease to be chronic
* Regulated hypertension
* Diabetes patients should have them blood sugar under 200 during therapy

Exclusion Criteria:

* Dementia
* Being a cancer patient receiving chemotherapy
* Epilepsy and a history of seizures
* Patient who has recently undergone surgery
* Pregnancy
* Delirium
* Bedridden

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | 2 weeks
  The Beck Depression Inventory is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Beck Depression Inventory is a 21-question multiple-choice self-report inventory The Beck Depression Inventory takes approximately 10 minutes to complete. The minimum score that can be obtained from the scale is 0 and the maximum score is 63 . Higher total scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Charlson Comorbidity Index | 2 weeks
  The Charlson Comorbidity Index is a method of categorizing comorbidities of patients. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.

OTHER OUTCOMES:
The Beck Anxiety Inventory | 2 weeks
  The Beck Anxiety Inventory is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The questions used in this measure ask about common symptoms of anxiety that the subject has had during the past week (including the day you take it) (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). It is designed for individuals who are of 17 years of age or older and takes 5 to 10 minutes to complete. The minimum score that can be obtained from the scale is 0 and the maximum score is 63.
MODIFIED FATIGUE IMPACT SCALE | 2 weeks
  The Modified Fatigue Impact Scale is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items. The minimum score that can be obtained from the scale is 0 and the maximum score is 84.
The Fatigue Severity Scale | 2 weeks
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer.
Ferrans and Powers quality of life index | 2 weeks
  The subjective perception of the level of happiness and satisfaction towards the different aspects of life is considered the main determinant in making a positive or negative judgment of the subjectively perceived quality of life. The current generic version of the Ferrans and Powers Quality of Life Index consists of 33 items in each part, which the subjects attribute scores in a satisfaction. The 33 items are distributed into the four dimensions (subscales): Health/functioning (13 items), Social and economic (8 items), Psychological/spiritual (7 items) and Family (5 items). The minimum score that can be obtained from the scale is 0 and the maximum score is 30.
Chest Circumference Measurement | 2 weeks
  Standing, it is measured by arms in abduction. It passes through the lower end of the scapula on the back and is measured at the level of the 4th rib.
Waist to Hip Ratio | 2 weeks
  It is the ratio of waist circumference to hip circumference. By measuring this value for scientific studies, it examines the risk level of potential health problems that individuals may encounter in the future. According to the studies of scientists, it shows quite accurate results about the risk of an individual having a health problem because it shows in which part of the body the excess weight is collected.
INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE | 2 weeks
  The International Physical Activity Questionnaires comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity. 1998 and was followed by extensive reliability and validity testing undertaken across 12 countries (14 sites) . Physical Activity level is determined in 3 categories

IPD SHARING:
Plan to Share IPD: No